CLINICAL TRIAL: NCT05937152
Title: CAT-Trial: CGRP Monoclonal Antibody for Treatment of Painful Diabetic Neuropathy: a Double-blind, Randomized, Placebo-controlled, International Multicenter, Phase II Clinical Trial
Brief Title: A Study of CGRP Monoclonal Antibody to Treat Diabetic Neuropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Narayan R. Kissoon, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 22-012864
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Eptinezumab Group (Experimental): Subjects diagnosed with diabetic polyneuropathy (DPN) will receive 2 infusions of eptinezumab during the 24 week-long placebo-controlled treatment period.
  Interventions: Drug: Eptinezumab
- Placebo Group (Placebo Comparator): Subjects diagnosed with diabetic polyneuropathy (DPN) will receive 2 infusions of placebo during the 24-week long placebo-controlled treatment period.
  Interventions: Drug: Placebo
- Open-label Eptinezumab Group (Experimental): At the end of the placebo-controlled treatment period, all participants will have the option to continue into the 24-week long active study treatment period and will receive 2 infusions of eptinezumab.
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — Intravenous (IV) infusion of 300 mg
  Arms: Eptinezumab Group; Open-label Eptinezumab Group
Drug: Placebo — Intravenous (IV) infusion of placebo (looks exactly like the study drug, but it contains no active ingredients)
  Arms: Placebo Group

SUMMARY:
The main purpose of this study is to compare the change in pain intensity during treatment with a CGRP monoclonal antibody (eptinezumab) compared with placebo treatment in patients with painful diabetic polyneuropathy (DPN).

DETAILED DESCRIPTION:
In neuropathy (nerve inflammation), which is seen in diabetes and other types of damage to the nerves, pain often occurs that can be difficult to treat. Some drugs have some effect on these pains, but unfortunately the treatment is not equally effective for all patients. It is not known why some patients achieve good pain relief with a given treatment. CGRP monoclonal antibody (eptinezumab) was originally developed as a drug for migraine and works by blocking molecules called CGRP that we, based on previous studies, play a major role in pain perception. Our previous studies have shown that patients with painful diabetic neuropathy (DPN) have increased incidence of the CGRP molecules in the skin precisely where patients experience pain compared to patients with painless DPN and healthy people without neuropathy. Eptinezumab is a Food and Drug Administration (FDA) approved drug for migraines, but it is not an approved drug for the treatment of DPN. The purpose of the trial is to investigate whether the treatment has an effect on the pain in the feet experienced by some patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of probable diabetic polyneuropathy, as defined by the Toronto consensus criteria and a TCNS > 5 or abnormal DPNCheck or abnormal NCS.
* Probable neuropathic pain as defined by the NeuPSIG guidelines.
* Symmetric distal pain worse in the distal lower extremities present for > 6 months.
* Average pain score on a NRS of ≥ 4 during the baseline week.

Exclusion Criteria:

* Prior or current use of a CGRP mAbs or CGRP antagonists.
* Opioid regimen other than stable low dose of Tramadol (maximum 200 mg/day).
* The patient has a lifetime history of psychosis, bipolar mania, or dementia. Patients with other psychiatric conditions whose symptoms are not controlled or who have not been adequately treated for a minimum of 6 months prior to screening are also excluded.
* Initiation of new neuropathic pain medications such as gabapentinoid medications (gabapentin, pregabalin) and/or capsaicin (Quetenza), botulinum toxin type A, serotonin/norepinephrine reuptake inhibitors (TCA or duloxetine or venlafaxine) 1 month prior to enrollment or for the duration of the randomized placebo-controlled phase of the study. Current and ongoing pain treatment will be allowed in stable dose (anticonvulsants, antidepressants, tramadol, topical treatments (excluding high dose capsaicin patch and botulinum toxin type A) (Paracetamol 1g and over-the-counter NSAIDS as needed up to four times daily are allowed as rescue medicine).
* Suspected cause of lower extremity pain of other causes than diabetes (e.g., chemotherapy, alcohol or drug misuse, vitamin deficiency, concomitant central nervous system pathology) or patients with pain that cannot be distinguished from their neuropathic pain in the feet due to diabetes.
* The patient has a history of clinically significant cardiovascular disease, including uncontrolled hypertension, ischaemia or thromboembolic events (for example, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism).
* The patient has a BMI ≥ 39 kg/m^2 at the screening visit.
* Peripheral arterial disease (PAD) defined as toe pressure < 40mmHg, no palpable foot pulses or clinical claudicatio intermittens.
* Chronic wounds.
* Planned larger surgery in the treatment period.
* Unable to understand Danish (Danish site only).
* All female subjects of childbearing potential must have negative result of a serum pregnancy test performed at screening. Subjects of childbearing potential must agree to use a medically approved form of birth control (abstinence, intrauterine device (IUD), oral contraception, barrier and spermicide or hormonal implant) throughout the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline, 24 weeks
  Weekly self-reported mean pain intensity (mean pain over the last 24 h recorded every morning in every fourth week in a diary) by the average numerical rating scale (NRS) on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
Change in Neuropathic Pain Severity | Baseline, week 12 and week 24
  Measured by the total score of Neuropathic Pain Scale (NPS) on a scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Pain relief at 12 weeks | 12 weeks
  Measured using a scale of complete, good, moderate, mild, none, worse
Pain relief at 24 weeks | 24 weeks
  Measured using a scale of complete, good, moderate, mild, none, worse

CONTACTS AND LOCATIONS:
Overall Officials: Narayan Kissoon, MD, Principal Investigator — Mayo Clinic
Locations (3):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States
- Denmark (2):
  - Steno Diabetes Center Aarhus, Aarhus
  - Steno Diabetes Center Copenhagen, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials